CLINICAL TRIAL: NCT05327972
Title: DEgenerative ROtator Cuff Disease and Botulinum TOXin: a Randomized Trial
Brief Title: DEgenerative ROtator Cuff Disease and Botulinum TOXin
Acronym: DEROTOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP210416
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Degenerative Rotator Cuff Disease
Keywords: Degenerative rotator cuff disease; Botulinum toxin; Clinical trial
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1- Botulinum toxin (Experimental): The investigational medicinal product is incobotulinumtoxinA (XEOMIN®).
  The dosage is:
  Two milliliters of a mixture comprised of XEOMIN® 100 U and saline solution 0.9% will be once injected in the supra-spinatus muscle using ultrasonography guidance.
  Interventions: Drug: The investigational medicinal product is incobotulinumtoxinA (XEOMIN®).
- 2- PLACEBO (Placebo Comparator): The placebo comparator represents a saline solution containing an inactive lyophilisate.
  The dosage is:
  Two milliliters of a saline solution containing an inactive lyophilisate will be once injected in the supra-spinatus muscle using ultrasonography guidance.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: The investigational medicinal product is incobotulinumtoxinA (XEOMIN®). — Two milliliters of a mixture comprised of XEOMIN® 100 U and saline solution 0.9% will be once injected in the supra-spinatus muscle using ultrasonography guidance.
  Arms: 1- Botulinum toxin
Other: PLACEBO — Two milliliters of a saline solution containing an inactive lyophilisate will be once injected in the supra-spinatus muscle using ultrasonography guidance.
  Arms: 2- PLACEBO

SUMMARY:
The aim of the study is to assess the effectiveness of botulinum toxin in persistent shoulder pain due to degenerative rotator cuff disease.

DETAILED DESCRIPTION:
Epidemiology:

degenerative rotator cuff disease ranks first in shoulder disorders and is the main cause of chronic shoulder pain in general practice and in rheumatology clinics. It can be responsible for persistent shoulder pain, functional limitation and greatly contributes to occupational disability.

The pathogenesis of rotator cuff disease:

involves tendon impingement and intrinsic tendinopathic abnormality (supra-spinatus, infra-spinatus, teres minor and sub-scapularis muscles). They include apoptosis of the tenocytes that is induced by mechanical constraints and by local hypoxia. The consequences are secondary inflammation and matrix alteration.

Current therapeutic approach:

The first-line recommended treatment for degenerative rotator cuff disease is conservative and includes level 1 and 2 oral analgesics; a short sequence of nonsteroidal anti-inflammatory drugs, if necessary; local injections of corticosteroids; and physiotherapy (low level of evidence). Surgery is a conditional later option.

Study hypothesis:

Reducing mechanical constraints on the supra-spinatus tendon by botulinum toxin may prevent load-induced apoptosis of the tenocytes and tear progression that is associated with clinical expression, and prevent local hypoxia. Furthermore, the muscle inactivity induced by botulinum toxin is not awaited to provide any clinically relevant functional alteration.

Aim of the study:

The primary objective of the study is to assess the effectiveness of botulinum toxin in persistent shoulder pain due to degenerative rotator cuff disease at one-month follow-up, using Shoulder Pain And Disability Index (SPADI) as outcome criterion.

The secondary objective is to assess the effectiveness of botulinum toxin in persistent shoulder pain due to degenerative rotator cuff disease, at three-month follow-up, using SPADI as outcome criterion and safety, the SPADI sub-scores pain and function at 3 months, global improvement perceived at 1 month and 3 months, drug consumption over the 3 months of follow-up, and treatment acceptability at 1 month and 3 months; as well as the tolerance at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* age > 40 years;
* pain duration > 1 month;
* pain intensity ≥ 40/100 on visual analog scale;
* SPADI ≥ 30/100;
* medication against pain stable at least 30 days before enrolment;
* pain with or without weakness during the Jobe manoeuver;
* ultrasonography within the 30 days, showing tendinopathy of the supra-spinatus, with or without tear;
* affiliation to health insurance Sécurité Sociale;
* ability to give consent, complete the weekly notebook (collection of drug treatments taken against pain);
* availability for the visits planned by the protocol;
* use of an effective method of contraception in women of childbearing potential, started at least 1 month before and lasting for at least 1 month after receiving study treatment.
* Negative urine test for women of childbearing age

Exclusion Criteria:

* reduced passive range of motion;
* antero-posterior instability;
* tendinous calcification;
* ultrasonography showing concomitant tear of the infra-spinatus or the subscapularis;
* corticosteroid injection within the previous 30 days;
* previous surgery of the shoulder;
* humeral fracture, inflammatory joint disease and neoplastic disorders;
* contraindication to XEOMIN® (allergy to XEOMIN® or any other botulinum toxin product);
* skin infection at the planned injection site;
* participation in another interventional research involving the human person (RIPH) during the 3 months of follow-up of the DEROTOX Research; participation in another RIPH will be possible beyond these 3 months;
* concomitant use of aminoglycosides, cyclosporine, aminoquinolines and spectinomycine;
* patients with a history of aspiration pneumonia and dysphagia;
* patients on anticoagulant therapy or on therapy that may have an anticoagulant effect;
* Patients with bleeding disorders;
* Patients with amyotrophic lateral sclerosis, myasthenia gravis or, Lambert-Eaton syndrome;
* Patients with other conditions causing peripheral neuromuscular dysfunction;
* In target muscles that show pronounced weakness or atrophy;
* Women of childbearing age who have not performed a urine pregnancy test and or who have a positive urine pregnancy test;
* in case of pregnancy, breastfeeding
* injection of botulinum toxin in the last 6 months
* vulnerable people (under legal protection, guardianship or curatorship)

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Total score of the Shoulder Pain And Disability Index at 1 month. 0 to 100; | 1 month
  Total score of the Shoulder Pain And Disability Index :
  Scale : 0 to 100, with higher score meaning worst outcome

SECONDARY OUTCOMES:
Sub-scores for pain and disability of the Shoulder Pain And Disability Index at 1 month and 3 months Total score of the Shoulder Pain And Disability Index at 3 months Safety at 1 week, 1 month and 3 months | week, 1 month and 3 months
  Sub-scores for pain and disability of the Shoulder Pain And Disability Index :
  Scale : 0 to 100, with higher score meaning worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johann MD BEAUDREUIL, PHD, Principal Investigator — Hôpital Lariboisière Fernand Widal
Locations (1):
- Hôpital LARIBOISIERE, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badley EM, Tennant A. Changing profile of joint disorders with age: findings from a postal survey of the population of Calderdale, West Yorkshire, United Kingdom. Ann Rheum Dis. 1992 Mar;51(3):366-71. doi: 10.1136/ard.51.3.366. PMID 1533506
- [Background] van der Heijden GJ. Shoulder disorders: a state-of-the-art review. Baillieres Best Pract Res Clin Rheumatol. 1999 Jun;13(2):287-309. doi: 10.1053/berh.1999.0021. PMID 10952865
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Bot SD, van der Waal JM, Terwee CB, van der Windt DA, Schellevis FG, Bouter LM, Dekker J. Incidence and prevalence of complaints of the neck and upper extremity in general practice. Ann Rheum Dis. 2005 Jan;64(1):118-23. doi: 10.1136/ard.2003.019349. PMID 15608309
- [Background] Linsell L, Dawson J, Zondervan K, Rose P, Randall T, Fitzpatrick R, Carr A. Prevalence and incidence of adults consulting for shoulder conditions in UK primary care; patterns of diagnosis and referral. Rheumatology (Oxford). 2006 Feb;45(2):215-21. doi: 10.1093/rheumatology/kei139. Epub 2005 Nov 1. PMID 16263781
- [Background] Hartvigsen J, Davidsen M, Hestbaek L, Sogaard K, Roos EM. Patterns of musculoskeletal pain in the population: a latent class analysis using a nationally representative interviewer-based survey of 4817 Danes. Eur J Pain. 2013 Mar;17(3):452-60. doi: 10.1002/j.1532-2149.2012.00225.x. Epub 2012 Oct 5. PMID 23042697
- [Background] Peters D, Davies P, Pietroni P. Musculoskeletal clinic in general practice: study of one year's referrals. Br J Gen Pract. 1994 Jan;44(378):25-9. PMID 8312034
- [Background] van der Windt DA, Koes BW, de Jong BA, Bouter LM. Shoulder disorders in general practice: incidence, patient characteristics, and management. Ann Rheum Dis. 1995 Dec;54(12):959-64. doi: 10.1136/ard.54.12.959. PMID 8546527
- [Background] Vecchio P, Kavanagh R, Hazleman BL, King RH. Shoulder pain in a community-based rheumatology clinic. Br J Rheumatol. 1995 May;34(5):440-2. doi: 10.1093/rheumatology/34.5.440. PMID 7788173
- [Background] Gartsman GM, Brinker MR, Khan M, Karahan M. Self-assessment of general health status in patients with five common shoulder conditions. J Shoulder Elbow Surg. 1998 May-Jun;7(3):228-37. doi: 10.1016/s1058-2746(98)90050-7. PMID 9658347
- [Background] Ostor AJ, Richards CA, Prevost AT, Speed CA, Hazleman BL. Diagnosis and relation to general health of shoulder disorders presenting to primary care. Rheumatology (Oxford). 2005 Jun;44(6):800-5. doi: 10.1093/rheumatology/keh598. Epub 2005 Mar 15. PMID 15769790
- [Background] Tekavec E, Joud A, Rittner R, Mikoczy Z, Nordander C, Petersson IF, Englund M. Population-based consultation patterns in patients with shoulder pain diagnoses. BMC Musculoskelet Disord. 2012 Nov 29;13:238. doi: 10.1186/1471-2474-13-238. PMID 23190941
- [Background] Virta L, Joranger P, Brox JI, Eriksson R. Costs of shoulder pain and resource use in primary health care: a cost-of-illness study in Sweden. BMC Musculoskelet Disord. 2012 Feb 10;13:17. doi: 10.1186/1471-2474-13-17. PMID 22325050
- [Background] Roquelaure Y, Ha C, Leclerc A, Touranchet A, Sauteron M, Melchior M, Imbernon E, Goldberg M. Epidemiologic surveillance of upper-extremity musculoskeletal disorders in the working population. Arthritis Rheum. 2006 Oct 15;55(5):765-78. doi: 10.1002/art.22222. PMID 17013824
- [Background] Wilson d'Almeida K, Godard C, Leclerc A, Lahon G. Sickness absence for upper limb disorders in a French company. Occup Med (Lond). 2008 Oct;58(7):506-8. doi: 10.1093/occmed/kqn084. Epub 2008 Jun 27. PMID 18587147
- [Background] Benson RT, McDonnell SM, Knowles HJ, Rees JL, Carr AJ, Hulley PA. Tendinopathy and tears of the rotator cuff are associated with hypoxia and apoptosis. J Bone Joint Surg Br. 2010 Mar;92(3):448-53. doi: 10.1302/0301-620X.92B3.23074. PMID 20190320
- [Background] Millar NL, Reilly JH, Kerr SC, Campbell AL, Little KJ, Leach WJ, Rooney BP, Murrell GA, McInnes IB. Hypoxia: a critical regulator of early human tendinopathy. Ann Rheum Dis. 2012 Feb;71(2):302-10. doi: 10.1136/ard.2011.154229. Epub 2011 Oct 4. PMID 21972243
- [Background] Yamaguchi K, Tetro AM, Blam O, Evanoff BA, Teefey SA, Middleton WD. Natural history of asymptomatic rotator cuff tears: a longitudinal analysis of asymptomatic tears detected sonographically. J Shoulder Elbow Surg. 2001 May-Jun;10(3):199-203. doi: 10.1067/mse.2001.113086. PMID 11408898
- [Background] Beaudreuil J, Dhenain M, Coudane H, Mlika-Cabanne N. Clinical practice guidelines for the surgical management of rotator cuff tears in adults. Orthop Traumatol Surg Res. 2010 Apr;96(2):175-9. doi: 10.1016/j.otsr.2010.02.002. PMID 20464793
- [Background] Page MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012224. doi: 10.1002/14651858.CD012224. PMID 27283590
- [Background] Placzek R, Drescher W, Deuretzbacher G, Hempfing A, Meiss AL. Treatment of chronic radial epicondylitis with botulinum toxin A. A double-blind, placebo-controlled, randomized multicenter study. J Bone Joint Surg Am. 2007 Feb;89(2):255-60. doi: 10.2106/JBJS.F.00401. PMID 17272437
- [Background] Wuelker N, Schmotzer H, Thren K, Korell M. Translation of the glenohumeral joint with simulated active elevation. Clin Orthop Relat Res. 1994 Dec;(309):193-200. PMID 7994959
- [Background] Collin P, Matsumura N, Ladermann A, Denard PJ, Walch G. Relationship between massive chronic rotator cuff tear pattern and loss of active shoulder range of motion. J Shoulder Elbow Surg. 2014 Aug;23(8):1195-202. doi: 10.1016/j.jse.2013.11.019. Epub 2014 Jan 14. PMID 24433628
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601
- [Background] Jobe FW, Moynes DR. Delineation of diagnostic criteria and a rehabilitation program for rotator cuff injuries. Am J Sports Med. 1982 Nov-Dec;10(6):336-9. doi: 10.1177/036354658201000602. PMID 7180952
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- See also: Haute Autorité de Santé. Clinical practice guidelines. Management of chronic painful shoulder without instability in adults. April 2005 — http://www.has-sante.fr
- See also: Rouvière H, Delmas A. Anatomie humaine, descriptive, topographique et fonctionnelle, tome 3 : membres, système nerveux central. 13ème édition. Paris : Masson ; 1991 — https://www.elsevier-masson.fr